CLINICAL TRIAL: NCT05719844
Title: Interest of an Attentional Evaluation by a Computerized Battery in the Management of Concussion in Young Rugby Players
Acronym: NeuropsyCor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOI 2021 VIDAL
Record Dates: First submitted 2023-01-17; First posted 2023-02-09 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-01

CONDITIONS: Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuropsychological tests (Experimental): The neuropsychological tests are computerized (TAP battery) or paper-and-pencil tests. They assess processing speed, short-term memory and auditory-verbal working memory capacity, episodic memory and selective attention.
  Interventions: Diagnostic Test: Neuropsychological tests

INTERVENTIONS:
Diagnostic Test: Neuropsychological tests — List of neuropsychological tests:
  * Matrix reasoning
  * D2-R
  * Coding
  * Symbol search
  * Digit span
  * Alertness (computerized TAP battery)
  * Divided Attention (computerized TAP battery)
  * Go / No go (computerized TAP battery)
  * Incompatibility (computerized TAP battery)
  * Working memory (computerized TAP battery)
  * 16-item Free and Cued Recall or Stories subtest of the Children Memory Scale (CMS) for children only (< 17 years old)
  * complex figure of the memory efficiency battery 144 or Word pairs of the Children Memory Scale for children only (< 17 years old)

SUMMARY:
The goal of this study is to test the ability of a computerized neuropsychological battery to identify attentional disorders resulting from a concussion occurring during the practice of rugby. Thirty young people with a concussion (11-25 years old) will take several neuropsychological tests. Researchers will compare their results with those of young athletes without concussion to see the effect of concussion.

DETAILED DESCRIPTION:
The objective is to carry out a complete neuropsychological assessment, detailing the attentional and executive aspects using the TAP computerized battery. In addition, various paper-and-pencil tests, standardized in French, more commonly used in the context of neuropsychological data related to concussions in athletes, will also be administered. These assess processing speed, short-term memory and auditory-verbal working memory capacity, episodic memory and selective attention. This preliminary study would make it possible to shed light on the links that may exist between performance in the various tests proposed and the characteristics inherent in the symptomatology of concussion. Furthermore, it seems relevant to compare the results of computerized tests with other paper-and-pencil tests but also with the performance of individuals who have no history of concussion with the practice of a non-contact sport.

The results of this study would make it possible in practice to have a neuropsychological assessment more specific to cerebral concussion, with a potentially reduced consultation time due to the use of more sensitive tools, and therefore, an earlier rehabilitative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients :
* concussion in the context of the practice of rugby
* French or reading French without help
* Controls :
* no concussion
* practicing a non-contact sport (athletics, rowing, badminton, capoeira, circus, running, crossfit, cycling, dancing, climbing, fencing, fitness, golf, gymnastics, bodybuilding, swimming, skating, Qi Gong, Taï chi, tennis, table tennis, shooting, trail running, volleyball, water polo) within a sports association
* age matched to patient (+/- 1 year)
* study level matched to patient (+/- 1 year)
* French or reading French without help

Exclusion Criteria:

* Patients :
* Legal protection measure
* Other neurological or psychiatric pathologies prior to concussion episodes
* Diagnosis of a neurodevelopmental disorder in childhood
* Score less than or equal to 5/19 on the "Matrix" subtest (intellectual retardation)
* Addictive behaviors
* Current major depressive disorder or treated with antidepressants or benzodiazepines for less than 3 months
* Severe visual or motor problems that may interfere with the performance of the tests
* Controls :
* Legal protection measure
* History of proven concussion
* Other neurological or psychiatric pathologies
* Diagnosis of a neurodevelopmental disorder in childhood
* Score less than or equal to 5/19 on the "Matrix" subtest (intellectual retardation)
* Addictive behaviors
* Current major depressive episode or treated with antidepressants or benzodiazepines for less than 3 months
* Severe visual or motor problems that may interfere with the performance of the tests

Ages: 11 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Alertness time | At inclusion
  Reaction time (ms) in the Alertness TAP test
Alertness error | At inclusion
  Number of errors in the Alertness TAP test
Divided Attention time | At inclusion
  Reaction time (ms) in the Divided Attention TAP test
Divided Attention error | At inclusion
  Number of errors in the Divided Attention TAP test
Go/No-go time | At inclusion
  Reaction time (ms) in the Go/No-go TAP test
Go/No-go error | At inclusion
  Number of errors in the Go/No-go TAP test
Incompatibility time | At inclusion
  Reaction time (ms) in the Incompatibility TAP test
Incompatibility error | At inclusion
  Number of errors in the Incompatibility TAP test
Working Memory time | At inclusion
  Reaction time (ms) in the Working Memory TAP test
Working Memory error | At inclusion
  Number of errors in the Working Memory TAP test

SECONDARY OUTCOMES:
Matrix reasoning | At inclusion
  Number of errors in Matrix reasoning test
Coding | At inclusion
  Number of errors in coding test
Symbol | At inclusion
  Number of errors symbol search test
Digit span | At inclusion
  Number of errors in digit span test
16-item free and cued recall | At inclusion
  Number of recall words in 16-item free and cued recall test
Complex figure | At inclusion
  Score in the complex figure of the memory efficient battery 144. Score is determined by the number of elements of the figure recalled.
Stories | At inclusion
  Number of errors in stories subtests of the Child Memory Scale (CMS)
Word pairs | At inclusion
  Number of errors in word pairs subtests of the Child Memory Scale (CMS)
D2-R error | At inclusion
  Number of errors in D2-R tests
D2-R time | At inclusion
  Time (in seconds) to complete the D2-R test
Sociodemographic data | At inclusion
  age and level of study of participants
Headaches | At inclusion
  Presence or absence of headaches
Amnesia | At inclusion
  Presence of anterograde or retrograde amnesia
SCAT | At inclusion
  Symptom severity score on the Sport Concussion Assessment Tool (SCAT), range 0-132 (minimum-maximum), a higher score representing a more severe concussion
Sleep | At inclusion
  Change in sleep (presence of hyper or insomnia)
Consciousness | At inclusion
  Loss of initial consciousness or not
Position | At inclusion
  Player position in the rugby team

CONTACTS AND LOCATIONS:
Overall Officials: Tiphaine Vidal, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France